CLINICAL TRIAL: NCT05383378
Title: A Multi-center, Phase 1b, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Efficacy of Si-544 in Adults With Atopic Dermatitis
Brief Title: A First-In-Human Study to Evaluate the Safety, Tolerability, and Efficacy of Si-544 in Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: selectION Therapeutics GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SEL-001; 2021-003061-35 (EudraCT Number)
Record Dates: First submitted 2022-05-04; First posted 2022-05-20 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Eczema; Neurodermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Neurodermatitis

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts, a single ascending dose (SAD) part, and a multiple ascending dose (MAD) part.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- si-544 (Experimental): The study consists of 2 parts, an SAD and an MAD part. In both parts, subjects will be treated in cohorts and will be randomized within each cohort to treatment with si-544 or placebo.
  Interventions: Drug: si-544
- Placebo (Placebo Comparator): The study consists of 2 parts, an SAD and an MAD part. In both parts, subjects will be treated in cohorts and will be randomized within each cohort to treatment with si-544 or placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: si-544 — Subcutaneous injection in the abdomen
  Arms: si-544
Drug: Placebo — Subcutaneous injection in the abdomen
  Arms: Placebo

SUMMARY:
This is a multi-center, Phase 1b, double-blind, placebo-controlled, SAD and MAD, first-in-human study in subjects with mild to severe AD receiving si-544. The study consists of 2 parts, an SAD and an MAD part. In both parts, subjects will be treated in cohorts and will be randomized within each cohort to treatment with si-544 or placebo. Initially, 2 sentinel subjects will be treated (randomized to placebo or si-544) in each cohort.

ELIGIBILITY:
SAD and MAD part

1. Subject has the capacity for consenting, was informed about the nature, the scope, and the relevance of the clinical study, voluntarily agrees in participation and in the study provisions, and duly signed the informed consent form approved by the ethics committee before any study-related procedure.
2. Men and women aged ≥18 to 75 years
3. Willing and able to adhere to the protocol requirements
4. {deleted}
5. Women of childbearing potential must:

   1. have a negative pregnancy test (blood) at Screening.
   2. agree to use, and be able to comply with, highly effective measures of contraceptive control (failure rate less than 1% per year when used consistently and correctly) without interruption, from Screening through 30 days after the last IMP treatment.

   Reliable methods for this study are:

   i. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal) ii. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) iii. intrauterine device iv. intrauterine hormone-releasing system v. bilateral tubal occlusion vi. vasectomized sexual partner (provided that the partner is the sole sexual partner of the woman of childbearing potential and has received medical assessment of the surgical success) vii. sexual abstinence (only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment) Abstinence is only accepted as true abstinence: when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods and withdrawal] is not an acceptable method of contraception).

   c. agree to abstain from breast feeding during the study participation and for 90 days after the last IMP treatment.

   Postmenopausal (no menses for at least 1 year without alternative medical cause) or surgically sterile women (tubal ligation, hysterectomy, or bilateral oophorectomy) may be enrolled.
6. Men must practice true abstinence or agree to use a condom during sexual contact with a pregnant woman or a woman of childbearing potential for at least 90 days after the last IMP treatment, even after undergoing a successful vasectomy.

   SAD part only
7. Clinical diagnosis of mild to severe AD

   MAD part only
8. Clinical diagnosis of mild to severe AD with a SCORAD ≥15

Exclusion Criteria:

SAD and MAD part

1. Change (ie, starting anew, change in frequency, or change in drug substance) in standard systemic and topical therapy, or in immunosuppressive drug therapy within 4 weeks before Screening (for biologics such as dupilumab, the therapy may not be changed within 12 weeks before Screening), as judged by the investigator
2. Known history of hypersensitivity to constituents or excipients in the pharmaceutical formulation of the IMP
3. Uncontrolled hypertension or uncontrolled diabetes
4. History of seizures
5. Presence or history of paresthesia or neuropathy
6. Clinically significant ECG abnormalities, as judged by the investigator
7. Clinically relevant hepatic, neurological, pulmonary, ophthalmological, endocrine, renal, or other major systemic disease, as judged by the investigator
8. Presence of acute infection within 7 days before Screening, as judged by the investigator
9. Known or active infection with Mycobacterium tuberculosis
10. Known or active infection with human immunodeficiency virus, hepatitis B virus, or hepatitis C virus
11. Vaccination within 2 weeks before Screening and/or planned vaccination during the SAD part or the treatment period of the MAD part
12. Pregnancy
13. Any finding or medical condition prohibiting the inclusion in the study, as judged by the investigator
14. Current or previous (within 4 weeks before Screening) participation in another clinical study with an investigational medicinal product or medical device
15. Known or suspected abuse of alcohol, drugs, or medicinal products
16. Employee of the sponsor, or employee, or relative of the investigator
17. Use of prohibited medication
18. Subjects committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
19. Legal incapacity or limited legal capacity

    MAD part
20. Previous participation in the SAD part of this study with IMP dosing within 3 months before the planned first dosing of the MAD part.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  AEs will be summarized and tabulated according to the primary system organ class and preferred term. Separate analyses will be conducted using severity, seriousness, and relationship to the IMP.
Adverse events (AEs) | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  AEs will be summarized and tabulated according to the primary system organ class and preferred term. Separate analyses will be conducted using severity, seriousness, and relationship to the IMP.
Change from Baseline in hematology parameter plateletes to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of hematology parameter platelets the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter plateletes to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of hematology parameter platelets the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter erythrocytes to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of hematology parameter erythrocytes the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter erythrocytes to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of hematology parameter erythrocytes the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter leukocytes to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of hematology parameter leukocytes the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter leukocytes to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of hematology parameter leukocytes the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter differential leukocyte count to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of hematology parameter differential leukocyte count the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter differential leukocyte count to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of hematology parameter differential leukocyte count the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter hemoglobin to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of hematology parameter hemoglobin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter hemoglobin to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of hematology parameter hemoglobin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter hematocrit to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of hematology parameter hematocrit the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter hematocrit to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of hematology parameter hematocrit the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter mean corpuscular volume to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of hematology parameter mean corpuscular volume the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter mean corpuscular volume to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of hematology parameter mean corpuscular volume the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter mean corpuscular hemoglobin to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of hematology parameter mean corpuscular hemoglobin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter mean corpuscular hemoglobin to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of hematology parameter mean corpuscular hemoglobin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection
Change from Baseline in hematology parameter mean corpuscular hemoglobin concentration to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of hematology parameter mean corpuscular hemoglobin concentration the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in hematology parameter mean corpuscular hemoglobin concentration to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of hematology parameter mean corpuscular hemoglobin concentration the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in alanine aminotransferase to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of alanine aminotransferase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in alanine aminotransferase to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of alanine aminotransferase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in aspartate aminotransferase to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of aspartate aminotransferase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in aspartate aminotransferase to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of aspartate aminotransferase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in gamma-glutamyl transferase to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of gamma-glutamyl transferase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in gamma-glutamyl transferase to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of gamma-glutamyl transferase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in alkaline phosphatase to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of alkaline phosphatase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in alkaline phosphatase to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of alkaline phosphatase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in total bilirubin to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of total bilirubin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in total bilirubin to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of total bilirubin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in unconjugated (indirect) bilirubin to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of unconjugated (indirect) bilirubin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in unconjugated (indirect) bilirubin to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of unconjugated (indirect) bilirubin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in conjugated (direct) bilirubin to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of conjugated (direct) bilirubin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in conjugated (direct) bilirubin to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of conjugated (direct) bilirubin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood urea nitrogen to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood urea nitrogen the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood urea nitrogen to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood urea nitrogen the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in creatinine to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of creatinine the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in creatinine to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of creatinine the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in uric acid to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of uric acid the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in uric acid to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of uric acid the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in estimated glomerular filtration rate to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of estimated glomerular filtration rate the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in estimated glomerular filtration rate to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of estimated glomerular filtration rate the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter sodium to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter sodium the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter sodium to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter sodium the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter potassium to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter potassium the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter potassium to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter potassium the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter magnesium to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter magnesium the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter magnesium to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter magnesium the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter chloride to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter chloride the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter chloride to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter chloride the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter inorganic phosphate to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter inorganic phosphate the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter inorganic phosphate to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter inorganic phosphate the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter calcium to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter calcium the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter calcium to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter calcium the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter creatine phosphokinase to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter creatine phosphokinase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter creatine phosphokinase to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter creatine phosphokinase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter amylase to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter amylase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter amylase to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter amylase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter lipase to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter lipase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter lipase to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter lipase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter total protein to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter total protein the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter total protein to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter total protein the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter albumin to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter albumin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter albumin to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter albumin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter glucose (non-fasting) to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter glucose (non-fasting) the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry parameter glucose (non-fasting) to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter glucose (non-fasting) the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry hemoglobin A1c to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter hemoglobin A1c the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry hemoglobin A1c to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter hemoglobin A1c the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry triglycerides to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter triglycerides the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry triglycerides to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter triglycerides the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry cholesterol to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter cholesterol the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry cholesterol to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter cholesterol the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry ferritin to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter ferritin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry ferritin to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter ferritin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry D-dimer to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter D-dimer the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry D-dimer to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter D-dimer the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry lactate dehydrogenase to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter lactate dehydrogenase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry lactate dehydrogenase to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter lactate dehydrogenase the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry C-reative protein to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood biochemistry parameter C-reactive protein the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood biochemistry C-reative protein to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood biochemistry parameter C-reactive protein the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood coagulation partial thromboplastin time to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood coagulation parameter partial thromboplastin time the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood coagulation partial thromboplastin time to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood coagulation parameter partial thromboplastin time the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood coagulation parameter prothrombin time to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood coagulation parameter prothrombin time the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood coagulation parameter prothrombin time to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood coagulation parameter prothrombin time the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood coagulation parameter international normalized ratio (INR) all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood coagulation parameter international normalized ratio (INR) the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood coagulation parameter international normalized ratio (INR) all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood coagulation parameter international normalized ratio (INR) the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter pH to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of urinalysis parameter pH the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter pH to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of urinalysis parameter pH the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter leukocytes to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of urinalysis parameter leukocytes the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter leukocytes to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of urinalysis parameter leukocytes the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter nitrites to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of urinalysis parameter nitrites the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter nitrites to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of urinalysis parameter nitrites the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter blood to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of urinalysis parameter blood the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter blood to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of urinalysis parameter blood the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter protein to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of urinalysis parameter protein the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter protein to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of urinalysis parameter protein the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter glucose to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of urinalysis parameter glucose the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter glucose to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of urinalysis parameter glucose the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter ketones to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of urinalysis parameter ketones the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter ketones to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of urinalysis parameter ketones the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter urobilinogen to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of urinalysis parameter urobilinogen the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter urobilinogen to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of urinalysis parameter urobilinogen the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter bilirubin to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of urinalysis parameter bilirubin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in urinalysis parameter bilirubin to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of urinalysis parameter bilirubin the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in 12-lead ECG parameter PR-interval to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of 12-lead ECG parameter PR-interval the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in 12-lead ECG parameter PR-interval to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of 12-lead ECG parameter PR-interval the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in 12-lead ECG parameter QRS-interval to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of 12-lead ECG parameter QRS-interval the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in 12-lead ECG parameter QRS-interval to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of 12-lead ECG parameter QRS-interval the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in 12-lead ECG parameter QT-interval to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of 12-lead ECG parameter QT-interval the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in 12-lead ECG parameter QT-interval to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of 12-lead ECG parameter QT-interval the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in 12-lead ECG parameter QTc[F]-interval to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of 12-lead ECG parameter QTc[F]-interval the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in 12-lead ECG parameter QTc[F]-interval to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of 12-lead ECG parameter QTc[F]-interval the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in peripheral oxygen saturation to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of peripheral oxygen saturation the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in peripheral oxygen saturation to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of peripheral oxygen saturation the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood pressure to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of blood pressure the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in blood pressure to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of blood pressure the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in heart rate to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of heart rate the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in heart rate to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of heart rate the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in respiration rate to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of respiration rate the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in respiration rate to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of respiration rate the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in body temperature to all assessments during the study | SAD part: Between Day 1 (IMP injection) and Day 8 (last visit)
  For the analyses of body temperature the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.
Change from Baseline in body temperature to all assessments during the study | MAD part: Between Day 1 (first IMP injection) and Day 106 (last visit)
  For the analyses of body temperature the absolute values, and changes from Baseline will be summarized for all assessed time points. Baseline is defined as the last assessment before IMP injection.

SECONDARY OUTCOMES:
SAD part: Plasma concentration of free si-544 in blood plasma at Day 1 | Day 1
  Blood collections up to 15 minutes before, and immediately, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, and 8 hours after IMP injection. The sampling window will be ±1 minute for ≤1 hour, ±5 minutes for 2 hours, ±15 minutes for 4 hours, and ±30 minutes for 8 hours post injection.
  Plasma concentration of free si-544 in blood plasma will be analyzed by descriptive statistics by treatment group.
MAD part: Plasma concentration of free si-544 in blood plasma at Days 1 and 25 | Day 1 and Day 25
  Blood collections up to 15 minutes before, and immediately, 5 minutes, 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, and 8 hours after IMP injection. The sampling window will be ±1 minute for ≤1 hour, ±5 minutes for 2 hours, ±15 minutes for 4 hours, and ±30 minutes for 8 hours post injection.
  Plasma concentration of free si-544 in blood plasma will be analyzed by descriptive statistics by treatment group and visit.
MAD part: Change from Baseline in number of T cells in peripheral blood at Day 29, and Weeks 8, 12, and 16 | Day 1, Day 29, Week 8, Week 12, and Week 16 (last visit)
  Blood sampling window on Day 1: up to 15 minutes before IMP injection.
MAD part: Change from Baseline in immunophenotyping of T-cell subsets at Day 29, and Weeks 8, 12, and 16 | Day 1, Day 29, Week 8, Week 12, and Week 16 (last visit)
  Blood sampling window on Day 1: up to 15 minutes before IMP injection.
MAD part: Change from Baseline in serum cytokine levels at Day 29, and Weeks 8, 12, and 16 | Day 1, Day 29, Week 8, Week 12, and Week 16 (last visit)
  Blood sampling window on Day 1: up to 15 minutes before IMP injection.
MAD part: Optional: Change from Baseline of expression levels of Kv1.3 vs KCa3.1 of effector memory T cells at Day 29, and Weeks 8, 12, and 16 | Day 1, Day 29, Week 8, Week 12, and Week 16 (last visit)
  Blood sampling window on Day 1: up to 15 minutes before IMP injection.
Change from Baseline in anti-drug antibodies against si-544 in serum at Day 29 | Day 1 and Day 29
  Blood sampling window on Day 1: up to 15 minutes before IMP injection.
Change from Baseline in inflamed areas using the body surface area index at Days 15 and 29, and Weeks 8, 12, and 16 | Day 1, Day 15, Day 29, Week 8, Week 12, and Week 16 (last visit)
  The body surface index will be used to assess the inflamed skin areas as percentage of the total body surface area (BSA). Percentage of BSA affected by AD with each body part accounted for by: head and neck: 9%, upper limbs: 9% each, lower limbs: 18% each, anterior trunk: 18%, back: 18%, and genitals: 1%. The score for each affected area is added up with the total possible (ie, all areas affected) score for being 100 (ie, 100% of BSA).
Change from Baseline in atopic dermatitis (AD) severity by SCOring AD (SCORAD) at Days 15 and 29, and Weeks 8, 12, and 16 | Day 1, Day 15, Day 29, Week 8, Week 12, and Week 16 (last visit)
  The AD severity assessment will be done by SCORing Atopic Dermatitis (SCORAD). SCORAD is a composite score of 3 components: (A) the BSA involved in AD, (B) the severity of 6 clinical signs, and (C) a subject-reported component assessing pruritus and sleep loss. The total score is calculated with a maximal total score of 103. A score <25 indicates mild, score 25-60 moderate, and score 61-103 severe AD.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Klostermann, Dr., Study Director — selectION Therapeutics GmbH
Locations (5):
- Germany (5):
  - selectION Clinical Trial Site, Berlin
  - selectION Clinical Trial Site, Hamburg
  - selectION Clinical Trial Site, Magdeburg
  - selectION Clinical Trial Site, Mainz
  - selectION Clinical Trial Site, Wuppertal

IPD SHARING:
Plan to Share IPD: No
Due to uncertainties in EU data protection legislation individual deidentified participant data are not shared. The main uncertainty is the concept of what "deidentified" means. It appears not to mean that the data set of a person is simply separated from the person's name. What additional operations have to be done appears to depend on technological capabilities to re-identify the persons associated with the data set. A common perception is that the technological capabilities for re-identification are permanently increasing. This could have the effect that public data sets that are regarded as deidentified now might become re-identifiable data sets in the future. Once this happens, the sponsor is no longer able to make the publication of the data sets un-happen. This could result in sanctioning by EU data protection authorities. The sponsor wants to avoid this.